CLINICAL TRIAL: NCT00138359
Title: The Effect of a Single Control Intervention in the T Solium Life Cycle
Brief Title: Mass Treatment T Solium Community Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-043
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-12

CONDITIONS: Intestinal Parasitism
Keywords: T solium, cysticercus, pig triquina, solitaria, intestinal parasites, Niclosamide, tapeworms, Taeniasis
MeSH Terms: conditions — Intestinal Diseases, Parasitic; Cestode Infections; Taeniasis | interventions — Niclosamide

INTERVENTIONS:
Drug: Niclosamide

SUMMARY:
Investigators from Cayetano Heredia University and Johns Hopkins University are doing this study. They want to see how people and pigs get infected with a parasite, called cysticercus (known as "pig triquina"). Cysticercus attacks the meat of pigs and the brains of people. In the intestine, the parasite is known as "solitaria". This study is to see how treatment in both people and pigs works to control the disease.

DETAILED DESCRIPTION:
This is a prospective intervention study to determine the efficacy and persistence of effect over time of a single, chemotherapy intervention in both the human and porcine population. Four villages will be selected to be treated against T solium adult (in humans) and larval forms (in pigs), and two villages will receive no intervention and will serve as control villages. Pigs in control villages will be followed during 3 months only, and then the human and porcine populations will receive the intervention treatment. The effect of this intervention will be measured by the prevalence of infection in pigs and parasitic burden of infected pigs at month 3, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

* All consenting individuals older than two years living in the study villages (6 endemic communities of the Northern coast of Peru)

Exclusion Criteria:

* Pregnancy (for antiparasitic treatment only).

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4200
Dates: Start 2004-12; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru